CLINICAL TRIAL: NCT04170998
Title: A Multicenter, Double-blind, Placebo-controlled, Randomized, Parallel, Phase III Clinical Trial to Evaluate the Efficacy and Safety of Evogliptin When Added to Ongoing Metformin and Dapagliflozin Combination Therapy in Patients With Type 2 Diabetes Who Have Inadequate Glycemic Control
Brief Title: Efficacy and Safety of Evogliptin When Added to Ongoing Metformin and Dapagliflozin Combination Therapy in Patients With Type 2 Diabetes Who Have Inadequate Glycemic Control
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DA1229_DMTD_III
Record Dates: First submitted 2019-11-13; First posted 2019-11-20 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — 4-(3-amino-4-(2,4,5-trifluorophenyl)butanoyl)-3-(tert-butoxymethyl)piperazin-2-one; dapagliflozin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evogliptin 5mg group (Experimental): Evogliptin 5mg/d + Dapagliflozin 10mg/d + Metformin ≥ 1000mg/d
  Interventions: Drug: Evogliptin 5mg; Drug: Dapagliflozin 10mg; Drug: Metformin ≥ 1000mg
- Evogliptin Placebo group (Placebo Comparator): Evogliptin Placebo + Dapagliflozin 10mg/d + Metformin ≥ 1000mg/d
  Interventions: Drug: Evogliptin Placebo; Drug: Dapagliflozin 10mg; Drug: Metformin ≥ 1000mg

INTERVENTIONS:
Drug: Evogliptin 5mg — Participants receive Evogliptin 5mg orally once a day
  Other Names: Suganon
  Arms: Evogliptin 5mg group
Drug: Evogliptin Placebo — Participants receive placebo to match Evogliptin 5mg orally once a day
  Other Names: Placebo
  Arms: Evogliptin Placebo group
Drug: Dapagliflozin 10mg — Participants receive Dapagliflozin orally once a day
  Other Names: Forxiga
Drug: Metformin ≥ 1000mg — Metformin are administered at the same dose and formulation.

SUMMARY:
A Multicenter, Double-blind, Placebo-controlled, Randomized, Parallel, Phase III Clinical Trial to Evaluate the Efficacy and Safety of Evogliptin When Added to Ongoing Metformin and Dapagliflozin Combination Therapy in Patients With Type 2 Diabetes Who Have Inadequate Glycemic Control

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type II diabetes mellitus aged 19 years or older
* Subjects who performed Dual therapies (complex allowed) for one of the following, along with meals and exercise therapy

  1. Subjects who are receiving metformin ≥ 1000 mg/d and dapagliflozin 10 mg/d at the same dose for at least 8 weeks prior to the screening visit
  2. Subjects who are receiving metformin ≥ 1000 mg/d and SGLT-2 inhibitor except for dapagliflozin at the same dose for at least 8 weeks prior to the screening visit
* Subjects with 7.0%≤HbA1c≤10.5% at screening visit
* Subjects with fasting plasma glucose ≤ 270mg/dL at screening visit
* Subjects with 18.5kg/m2≤BMI≤40kg/m2 at screening visit

Exclusion Criteria:

* Patients with type 1 diabetes, secondary diabetes, gestational diabetes, diabetic ketoacidosis, diabetic coma, pre-coma, lactic acidosis, and acute or chronic metabolic acidosis
* patients with Hypopituitarism or adrenal insufficiency, pulmonary infarction, severe pulmonary dysfunction and other hypoxemia
* Patients with severe infectious disease or severe traumatic systemic disorders
* End stage renal disease or dialysis patients
* Patients with Galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption
* Subjects with Liver cirrhosis, chronic active hepatitis B or C, cholecystitis, acromegaly, asthma or major skin allergies

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2021-12-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c (%) After 24 weeks | 24 weeks

SECONDARY OUTCOMES:
Change from baseline in FPG(mg/dL) After 24 weeks | 24 weeks
Change from baseline in HbA1c response rate(<7.0% ,<6.5%) After 24 weeks | 24 weeks
Change from baseline in 7-point SMBG After 24 weeks | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul St, Mary's Hospital,The Catholic University of Korea, Seoul, South Korea

REFERENCES:
- [Derived] Moon JS, Park IR, Kim HJ, Chung CH, Won KC, Han KA, Park CY, Won JC, Kim DJ, Koh GP, Kim ES, Yu JM, Hong EG, Lee CB, Yoon KH. Efficacy and Safety of Evogliptin Add-on Therapy to Dapagliflozin/Metformin Combinations in Patients with Poorly Controlled Type 2 Diabetes Mellitus: A 24-Week Multicenter Randomized Placebo-Controlled Parallel-Design Phase-3 Trial with a 28-Week Extension. Diabetes Metab J. 2023 Nov;47(6):808-817. doi: 10.4093/dmj.2022.0387. Epub 2023 Sep 26. PMID 37750183